CLINICAL TRIAL: NCT00216047
Title: A Phase I/II Study of PTK787 in Combination With Trastuzumab in Patients With Newly Diagnosed HER2 Overexpressing Locally Recurrent or Metastatic Breast Cancer: Hoosier Oncology Group Trial BRE04-80
Brief Title: PTK787 + Trastuzumab for HER2 Overexpressing Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low patient enrollment; toxicities
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Walther Cancer Institute (Other)
Responsible Party: Principal Investigator, Kathy Miller, MD, Professor, IU School of Medicine, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG BRE04-80
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — vatalanib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group Assignment (Experimental): Trastuzumab + PTK787 for HER2 positive patients
  Interventions: Drug: PTK787; Drug: Trastuzumab

INTERVENTIONS:
Drug: PTK787 — PTK787 daily
Drug: Trastuzumab — Trastuzumab 4 mg/kg IV week 1, followed by 2 mg/kg weekly with disease evaluation every other cycle*

SUMMARY:
HER2 gene amplification increases VEGF production in breast cancers; combined inhibition of HER2 and VEGF enhances response in xenograft models. The upregulation of VEGF in HER2-overexpressing breast cancers may contribute to the aggressive phenotype observed in HER2-positive breast cancer. New therapeutics targeting VEGF and/or its receptors may enhance the efficacy of trastuzumab monotherapy.

This trial will investigate the safety and efficacy of combined HER2 and VEGF inhibition.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

PTK787 daily plus trastuzumab 4 mg/kg IV week 1, followed by 2 mg/kg weekly with disease evaluation every other cycle.

Patients may continue treatment until disease progression or toxicity intervenes.

Performance Status: ECOG 0 or 1

Life Expectancy: Not specified

Hematopoietic:

* ANC > 1500 mm3
* Platelets > 100,000 mm3
* Hemoglobin > 9 g/dL
* PTT and INR < 1.5 x ULN

Hepatic:

* ALT and AST < 3 x ULN (< 5 x ULN in patients with known liver metastases)
* Alkaline phosphatase < 2.5 x ULN
* Serum bilirubin < 1.5 x ULN

Renal:

* Serum creatinine < 1.5 x ULN
* Proteinuria < 1+ by dipstick OR total urinary protein < 500 mg/24 hours with measured creatinine clearance (CrCl) ≥ 50 mL/min

Cardiovascular:

* No clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 6 months.
* LVEF > LLN by MUGA or ECHO (obtained within 28 days prior to being registered for protocol therapy)

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of breast cancer with evidence of measurable (1) unresectable, locally recurrent, or (2) metastatic disease. Locally recurrent disease must not be amenable to resection OR radiation with curative intent.
* Patient's disease may not involve more than 3 metastatic sites. In addition, patient may not be symptomatic from pulmonary metastasis or have liver metastasis involving > 50% of parenchyma.
* HER2 gene amplification by FISH. HER protein overexpression by immunohistochemistry will not be sufficient for entry.
* Negative pregnancy test

Exclusion Criteria:

* No prior cytotoxic chemotherapy or trastuzumab for locally recurrent or metastatic disease.
* No prior treatment with any VEGF inhibiting agents
* No history or presence of central nervous system (CNS) disease.
* No other forms of cancer therapy including radiation, chemotherapy and hormonal therapy within 21 days prior to being registered for protocol therapy.
* No major surgery within 28 days prior to being registered for protocol therapy.
* No uncontrolled hypertension (SBP > 170, DBP > 90), history of labile hypertension or history of poor compliance with antihypertensive therapy.
* No requirement for therapeutic anticoagulation, regular aspirin (> 325 mg/day) or NSAID use.
* No current breast feeding.
* No impairment of gastrointestinal (GI) function that may significantly alter the absorption of PTK787.
* No evidence of other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Phase I Cohorts: | 18 months
The primary objective is to ensure the safety and tolerability of the combination of Trastuzumab and PTK787, | 18 months
Phase II Cohorts: | 18 months
To assess response rate of PTK787 combined with trastuzumab in patients with newly diagnosed HER2 overexpressing | 18 months

SECONDARY OUTCOMES:
Phase II Cohorts: | 12 months
To assess the safety and tolerability of PTK787 combined with trastuzumab | 12 months
To assess the time to progression and clinical benefit of PTK787 combined with trastuzumab | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (8):
- United States (8):
  - Elkhart Clinic, Elkhart, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana

REFERENCES:
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/